CLINICAL TRIAL: NCT04035174
Title: Evaluation of the Diagnosis Performances of DEC LTS-2 Skin Patch for Onchocerciasis in Central Africa
Acronym: EOLoa
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study site was changed to another countr
Sponsor: Center for Research on Filariasis and Other Tropical Diseases, Cameroon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: C18-56
Record Dates: First submitted 2019-07-25; First posted 2019-07-29 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Onchocerciasis; Loiasis; Diagnoses Disease; Neglected Diseases
Keywords: Health Public
MeSH Terms: conditions — Onchocerciasis; Loiasis; Neglected Diseases

STUDY DESIGN:
Intervention Model Description: Each participant will have both a LTS-2 patch applied on the skin and a skin snip performed.
Who Masked: Outcomes Assessor
Masking Description: Results from LTS-2 patch will be immediately known by both participant and investigators ; but results from skin snips will be masked both for participant and investigators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LTS-2 DEC patch (Experimental): This is a transdermal device with diethylcarbamazine (DEC) applied directly on the skin. The reading will be done 24 hours after.
  Interventions: Diagnostic Test: LTS-2 DEC patch; Diagnostic Test: Skin snips
- Skin snip (Active Comparator): A skin snip will be performed using a 2 mm Holth corneoscleral's punch. Once done, the microfilariae of Onchocerca volvulus will be counted with a microscope.
  Interventions: Diagnostic Test: LTS-2 DEC patch; Diagnostic Test: Skin snips

INTERVENTIONS:
Diagnostic Test: LTS-2 DEC patch — After 24 hours, the patch will be removed, and then the reaction of the skin under the device will be assessed : no reaction, weak reaction (< 50% skin surface under the patch), medium reaction (> 50% skin surface under the patch), and important reaction (reaction on all the surface of the skin under the patch).
Diagnostic Test: Skin snips — Regarding skin snips, a reading will be done at 24 hours after incubation of the skin in saline serum during 24 hours.

SUMMARY:
This study aims at evaluating the diagnosis performances of the LTS-2 DEC patch for onchocerciasis compared to the gold standard which are the skin snips. This study will be conducted in Cameroon in two different areas : Ngog-Mapubi and Bafia Health Districts (one area only endemic for onchocerciasis, and one area endemic for both loiasis and onchocerciasis).

ELIGIBILITY:
Inclusion Criteria:

* All voluntary adults

Exclusion Criteria:

* General acute infection (temperature ≥ 38,5°C)
* Impaired general condition
* Ivermectin taken in the 6 last months
* Known allergies to one of the component of the patch
* Dermatological acute infection (bacterial, atopic, prurigo, or zona)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2022-10-30 (Estimated); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Tolerability of the patch | 24 hours
  Proportion of individuals having developed a generalized Mazzotti's reaction
Feasibility of the patch | 24 hours
  Proportion of individuals for whom the patches are spontaneously removed from the skin during the 24 hours.

SECONDARY OUTCOMES:
Diagnosis performances | 24 hours
  Assessment of the sensibility, specificity, and predictive values of the LTS-2 DEC patch compared to the results from the skin snips.
Loiasis and cross-reactivity assessment | 24 hours
  Loiasis impact of the diagnosis performances of the LTS-2 DEC patch. Loiasis will be assessed with thick blood smears and a microscopic examination ; and with PCR in the skin snips
Semi-quantitative scoring of the LTS-2 DEC patch results | 24 hours
  Relationship between the number of microfilariae of O. volvulus and the skin reaction under the patch (0 no reaction, 1: < 50% of the skin under the patch, 2: >50% of the skin under the patch, and 3: reaction under all the skin surface of the patch)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Recherche sur les filarioses et autres maladies tropicales (CRFilMT), Yaoundé, Cameroon

IPD SHARING:
Plan to Share IPD: Yes